CLINICAL TRIAL: NCT03874208
Title: Prediction for Coma Recovery in ICU With Comaweb: a Validation Study
Brief Title: Prediction for Coma Recovery With Comaweb
Acronym: COMASCORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D20180112; 2018-A02190-55 (Other: IDRCB number)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2019-02

CONDITIONS: Brain Injury, Coma; Cardiac Arrest (CA); Traumatic Brain Injury (TBI); Aneurysmal Subarachnoid Hemorrhages (aSAH)
Keywords: Outcome prediction; Disorders of Consciousness; Coma,; MRI; Brain injury
MeSH Terms: conditions — Brain Injuries; Coma; Heart Arrest; Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Consciousness Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Other): To assess the predictive accuracy of comaScore evaluated in the day 7 - day 45 period post brain injury to predict unfavorable outcome at 1-year after the first insult in patients admitted in ICU after CA, TBI and aSAH, that remain comatose at least 7 days after brain injury.
  Interventions: Other: MRI sequence
- Test group (Other): MRI calibration in each center : test protocol compliance, data transfer procedures and quality of the MRI sequences
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI sequence — An additional sequence to conventional MRI exam (Diffusion tensor imaging) lasting less than 10 min (depending on the MR scanner type and sequence used).
  Arms: Patient group
Other: MRI — MRI exam
  Arms: Test group

SUMMARY:
The general objective of the comaScore project is to provide an external validation of the accuracy of the comaScore, a score derived from magnetic resonance imaging (MRI), to predict 1 year outcome of patients unresponsive to simple orders after traumatic brain injury (TBI), aneurysmal subarachnoid hemorrhages (aSAH) and cardiac arrest (CA) in the day 7 - day 45 period post brain injury.

DETAILED DESCRIPTION:
The general objective of the comaScore project is to provide an external validation of the accuracy of the comaScore, a score derived from magnetic resonance imaging (MRI), to predict 1 year outcome of patients unresponsive to simple orders after traumatic brain injury (TBI), aneurysmal subarachnoid hemorrhages (aSAH) and cardiac arrest (CA) in the day 7 - day 45 period post brain injury. As recent studies reported late awakeners cases, even in cardiac arrest and, in contrary, that around 10% of patients with acute brain injury remain with permanent disorders of consciousness (DOC), the need of reliable prognosis tool at the early phase, while the patient is still in the ICU, is critical. ComaScore, based on the quantitative analysis of diffusion tensor imaging, was developed from a derivation cohort of 506 patients. It is much more performing than existing tools (IMPACT, OHCA) in this respect.

This study aims to prospectively validate the predictive accuracy of comaScore to predict unfavorable outcome at 1-year after the first insult, in an independent sample (external validation). Unfavorable outcome is defined as a Glascow Outcome Scale Extended (GOSE) of 1 to 3. This scale ranges from 1 to 8. Scores of 1 to 3 correspond to death, vegetative state, minimally conscious state or bedridden.

ELIGIBILITY:
Patient Inclusion criteria

1. Male or female subject of 18 years old or above
2. Affiliated to a social security system excluding "Aide Médicale d'État (AME)"
3. Hospitalized in an intensive care unit and requiring mechanical ventilation after TBI, aSAH or CA
4. Absence of response to simple orders not explained by sedation alone at inclusion
5. Patient within 7 to 45 days after onset of TBI, aSAH or CA
6. Scheduled MRI within 5 days after inclusion
7. Written informed consent to participate in the study must be obtained proxy/legal representative.

Patient non-inclusion criteria

1. MRI unavailability between day 7 and day 45 after brain injury
2. Origin of coma other than CA, TBI or aSAH
3. Pre-existing serious brain disease prior to coma status
4. Contra-indication to perform MRI
5. Subject protected by the law (curatorship or tutorship)

Patient secondary exclusion criteria

1. Consciousness recovery before MRI exam
2. Contra-indication to perform MRI (appeared / discovered after inclusion)

Healthy controls Inclusion criteria

1. Male or female subject from 18 to 65 years
2. Affiliated to a social security system excluding "Aide Médicale d'État (AME)".
3. No history of previous brain disease
4. No contra-indication to perform an MRI.
5. No pregnancy
6. Voluntarily agrees to participate by providing written informed consent

Healthy controls Non-Inclusion criteria

1. Subject protected by the law (curatorship or tutorship)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 611 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
The unfavorable outcome | 1 year after the initial brain injury
  The unfavorable outcome is defined as a Glascow Outcome Scale Extended (GOSE) of 1 to 3. This scale ranges from 1 to 8. Scores of 1 to 3 correspond to death, vegetative state, minimally conscious state or bedridden.

SECONDARY OUTCOMES:
Time-window-specific performances of the Comascore evaluation | day 7 to 15, day 16 to 25, day 26 to 35 or day 36 to 45
  To assess the impact of time from brain injury to MRI allowing to calculate comaScore on the predictive accuracy of comaScore (4 periods will be determined
Etiology-specific performances of the Comascore evaluation after cardiac arrest | 1 year after the initial brain injury
  " To assess the predictive accuracy of comaScore evaluated in the day 7 - day 45 period post brain injury to predict unfavorable outcome at 1-year after the first insult in patients admitted in ICU after CA or TBI or sSAH, that remain unresponsive to simple orders at least 7 days after brain injury."
Etiology-specific performances of the Comascore evaluation after traumatic brain injury | 1 year after the initial brain injury
  " To assess the predictive accuracy of comaScore evaluated in the day 7 - day 45 period post brain injury to predict unfavorable outcome at 1-year after the first insult in patients admitted in ICU after CA or TBI or sSAH, that remain unresponsive to simple orders at least 7 days after brain injury."
Etiology-specific performances of the Comascore evaluation after aneurysmal subarachnoid hemorrhages | 1 year after the initial brain injury
  " To assess the predictive accuracy of comaScore evaluated in the day 7 - day 45 period post brain injury to predict unfavorable outcome at 1-year after the first insult in patients admitted in ICU after CA or TBI or sSAH, that remain unresponsive to simple orders at least 7 days after brain injury."
Comparison between COMASCORE and OHCA score after cardiac arrest | 1 year after the initial brain injury
  To test the statistical difference in predictive accuracy between comaScore evaluated in the day 7 - day 45 period post brain injury and OHCA or IMPACT or WFNS score to predict unfavorable outcome at 1-year after the first insult in patients admitted in ICU after CA or TBI or aSAH, respectively, that remain unresponsive to simple orders at least 7 days after brain injury.
Comparison between COMASCORE and IMPACT score after traumatic brain injury | 1 year after the initial brain injury
  To test the statistical difference in predictive accuracy between comaScore evaluated in the day 7 - day 45 period post brain injury and OHCA or IMPACT or WFNS score to predict unfavorable outcome at 1-year after the first insult in patients admitted in ICU after CA or TBI or aSAH, respectively, that remain unresponsive to simple orders at least 7 days after brain injury.
Comparison between COMASCORE and WFNS score after aneurysmal subarachnoid hemorrhages | 1 year after the initial brain injury
  To test the statistical difference in predictive accuracy between comaScore evaluated in the day 7 - day 45 period post brain injury and OHCA or IMPACT or WFNS score to predict unfavorable outcome at 1-year after the first insult in patients admitted in ICU after CA or TBI or aSAH, respectively, that remain unresponsive to simple orders at least 7 days after brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Puybasset Louis, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre Hospitalier Saint-Jean, Perpignan, France